CLINICAL TRIAL: NCT03646474
Title: Evaluation of the Efficacy & Safety of a Single Dose Tranexamic Acid in Reducing Blood Loss During Cytoreductive Surgery and HIPEC
Brief Title: Single Dose Tranexamic Acid in Reducing Blood Loss During Cytoreductive Surgery and HIPEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Assisstant professor of Anesthesia ICU and pain Relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201617027.2p
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Cytoreductive Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tranexamic acid group (Active Comparator)
  Interventions: Drug: tranexamic Acid infusion
- placebo group (Placebo Comparator)
  Interventions: Drug: saline infusion

INTERVENTIONS:
Drug: tranexamic Acid infusion — The tranexamic Acid group will receive an intravenous bolus of (10 mg/kg) in 100 ml of normal saline over 20 minutes after induction of anesthesia and before surgical incision.
  Arms: tranexamic acid group
Drug: saline infusion — In the placebogroup, patients will receive a placebo of 100 mL 0.9% normal saline.
  Arms: placebo group

SUMMARY:
The Tranexamic Acid group will receive an intravenous bolus of (10 mg/kg) in 100 ml of normal saline over 20 minutes after induction of anesthesia and before surgical incision. In the control group, patients will receive a placebo of 100 mL 0.9% normal saline. The primary endpoint is reduction in blood loss, while the secondary endpoint was the number of patients needing transfusion and occurrence of postoperative thrombotic complications (myocardial infarction, stroke, pulmonary embolism, renal failure, or bowel infarction) within 30 days after surgery.

ELIGIBILITY:
Inclusion criteria

* ASA 1 and ASA 2 patients scheduled for colorectal cancer surgery.
* Age above 18 years & less than 65 years.

Exclusion criteria:

* Thrombophilia or any bleeding disorder.
* Previous or active thromboembolic disease.
* Family history of thromboembolism.
* Known Allergy to TA.
* Liver dysfunction.
* Preexisting renal dysfunction (serum creatinine >1.2 mg/dL).
* Coronary stent insertion within a year prior to operation.
* Cardiovascular problem (e.g., myocardial infarction, atrial fibrillation, angina, heart failure),
* Lifelong warfarin therapy for thromboembolism prophylaxis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
change in blood loss | 1st 24 hours.
  Blood loss will be calculated (volume estimated as the blood remaining in sponges and drapes and the volume in suction bottles during surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo University, Cairo, Egypt